CLINICAL TRIAL: NCT01382225
Title: A Phase 3 Multicenter, Randomized, Controlled, Double-Masked Study of Safety and Efficacy of Sodium Hyaluronate Ophthalmic Solution, 0.18% in Dry Eye Syndrome
Brief Title: Sodium Hyaluronate Ophthalmic Solution, 0.18% for Treatment of Dry Eye Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-09-045
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Results first posted 2013-07-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-05

CONDITIONS: Dry Eye Syndrome
Keywords: Dry eyes; Ocular discomfort
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Hyaluronate (Experimental): Sodium Hyaluronate Ophthalmic Solution, 0.18%, 1-2 drops instilled in each eye 3-6 times a day for 14 days
  Interventions: Drug: Sodium Hyaluronate Ophthalmic Solution, 0.18%
- Vehicle (Placebo Comparator): Inactive ingredients, 1-2 drops instilled in each eye 3-6 times a day for 14 days
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Sodium Hyaluronate Ophthalmic Solution, 0.18%
  Arms: Sodium Hyaluronate
Other: Vehicle — Inactive ingredients used as run-in and placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study was to determine if Sodium Hyaluronate, 0.18% is effective in treating the signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of dry eyes for at least 3 months.
* Ocular discomfort due to dry eyes.
* Presence of corneal and conjunctival staining.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Contact lens wear within 1 week before Screening and during the study.
* Ocular surgery (of any type, including laser surgery) or ocular trauma within the 4 months prior to Screening.
* Punctal plugs or punctal occlusion initiated within 3 months of screening
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1936 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michela Montecchi-Palmer, BS, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 56 investigative sites in the United States.
Pre-assignment Details: Of the 1936 subjects enrolled, 268 did not qualify for vehicle run-in and were exited as screen failures. Of the 1668 subjects receiving vehicle run-in, 214 did not qualify for randomization and were exited as screen failures. This reporting group includes the 1454 subjects randomized to receive treatment at Baseline Visit (Day 0).
Groups:
- Sodium Hyaluronate: Run-in, followed by Sodium Hyaluronate Ophthalmic Solution, 0.18%, 1-2 drops instilled in each eye 3-6 times a day for 14 days
- Vehicle: Run-in, followed by Vehicle, 1-2 drops instilled in each eye 3-6 times a day for 14 days
Period: Overall Study
Arm/Group | Sodium Hyaluronate | Vehicle
Started | 725 | 729
Completed | 711 | 722
Not Completed | 14 | 7
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Subject Withdrew Consent | 5 | 2
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Population: Of the 1454 subjects randomized, 4 withdrew participation prior to exposure to test article. This reporting group includes the 1450 subjects exposed to test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Hyaluronate | Vehicle | Total
Number analyzed (Participants) | 723 | 727 | 1450
Age, Customized [Number; unit: participants]
  18-64 years | 402 | 392 | 794
  ≥65 years | 321 | 335 | 656
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 590 | 594 | 1184
  Male | 133 | 133 | 266
Region of Enrollment [Number; unit: participants]
  United States | 723 | 727 | 1450

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lissamine Green Staining (LGS) Total Score at Day 7
Description: The investigator instilled an ophthalmic dye on the eye and rated staining in three areas (cornea, nasal, and temporal conjunctiva). Staining was rated on a 5-point scale from 0 to 4 (0=0% to 4=>45%). The LGS Total Score (0-12) is the sum of the three individual ratings. A more negative change indicates a greater amount of improvement.
Time Frame: Baseline, Day 7
Population: Modified Intent-to-Treat (mITT): The set of all randomized subjects who received at least one administration of the allocated product, had baseline efficacy measurement, had at least 1 post-baseline measurement and received the correct formulation of the lissamine green solution.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Vehicle: Vehicle, 1-2 drops instilled in each eye 3-6 times a day for 14 days
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Units on a scale
  Baseline | 4.9 (2.2) | 4.8 (2.1)
  Change from Baseline at Day 7 | -0.8 (1.8) | -0.7 (1.6)

2. Primary Outcome: Change From Baseline in Global Symptom Frequency (GSF) Total Score at Day 7
Description: The subject completed a questionnaire and rated the frequency of five common dry eye symptoms. Frequency was rated on a 4-point scale from 0 to 3 (0=never to 3=constantly). The GSF Total Score (0-15) is the sum of the five individual ratings. A more negative change indicates a greater amount of improvement.
Time Frame: Baseline, Day 7
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Units on a scale
  Baseline | 8.9 (2.3) | 9.1 (2.3)
  Change from Baseline at Day 7 | -1.6 (2.6) | -1.3 (2.4)

3. Secondary Outcome: Change From Baseline in LGS Total Score at Day 14
Description: as for outcome 1
Time Frame: Baseline, Day 14
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Units on a scale
  Baseline | 4.9 (2.2) | 4.8 (2.1)
  Change from Baseline at Day 14 | -1.2 (2.0) | -1.0 (1.8)

4. Secondary Outcome: Change From Baseline in GSF Total Score at Day 14
Description: as for outcome 2
Time Frame: Baseline, Day 14
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Units on a scale
  Baseline | 8.9 (2.3) | 9.1 (2.3)
  Change from Baseline at Day 14 | -2.3 (2.8) | -2.2 (2.8)

5. Secondary Outcome: Percentage Change From Baseline in Corneal Fluorescein Staining (CFS) Total Score
Description: The investigator instilled an ophthalmic dye on the eye and rated corneal staining by type, extent/surface area, and depth. Each staining was rated on a 5-point scale from 0 to 4 (0=no staining/0% to 4=patch/>45%/immediate diffuse stromal glow). The CFS Total Score (0-12) is the sum of the three individual ratings. A more negative percentage change indicates a greater amount of improvement.
Time Frame: Baseline, up to Day 14
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Percent change
  Baseline | 4.9 (2.1) | 4.8 (2.0)
  Change from Baseline at Day 7 | -10.0 (40.3) | -10.4 (36.9)
  Change from Baseline at Day 14 | -19.3 (46.6) | -16.1 (44.1)

6. Secondary Outcome: Percentage Change From Baseline in Schirmer I Score
Description: The investigator placed a paper strip on the eye under the lower lid and left it in place for 5 minutes. The Schirmer I Score was the length of the strip wetted by the tears (0-35 millimeters). A more positive percentage change indicates a greater amount of improvement.
Time Frame: Baseline, up to Day 14
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Percent change
  Baseline | 9.7 (8.6) | 10.1 (8.5)
  Change from Baseline at Day 7 | 52.1 (195.2) | 40.6 (139.8)
  Change from Baseline at Day 14 | 60.3 (273.2) | 47.0 (170.7)

7. Secondary Outcome: Percentage Change From Baseline in Global Symptom Intensity (GSI) Total Score
Description: The subject completed a questionnaire and rated the intensity of five common dry eye symptoms. Intensity was rated on a visual analog scale from 0-100 (0=no symptoms to 100=severe symptoms). The GSI Total Score (0 to 500) is the sum of the five individual ratings. A more negative percentage change indicates a greater amount of improvement.
Time Frame: Baseline, up to Day 14
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Percent change
  Baseline | 294.2 (80.8) | 295.8 (82.5)
  Change from Baseline at Day 7 | -18.9 (34.1) | -15.4 (34.5)
  Change from Baseline at Day 14 | -31.6 (37.7) | -26.9 (38.4)

8. Secondary Outcome: Percentage Change From Baseline in Global Symptom Composite Index (GSCI) Score
Description: For each of 5 common dry eye symptoms, the frequency (0-3) and intensity (0-100) scores were multiplied to obtain the symptom score (0-300). The 5 symptom scores were summed to obtain the Global Symptom Composite Index Score (0-1500). A more negative percentage change indicates a greater amount of improvement.
Time Frame: Baseline, up to Day 14
Population: Modified Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Percentage change
  Baseline | 594.8 (249.9) | 608.4 (258.0)
  Change from Baseline at Day 7 | -26.1 (43.6) | -22.4 (43.2)
  Change from Baseline at Day 14 | -40.1 (44.9) | -36.3 (44.4)

9. Secondary Outcome: Proportion of Improved Scores on the Global Impact on Dry Eye Syndrome on Daily Life (GIDL) Rating
Description: The subject was asked on a questionnaire, "Please consider how your dry eyes feel when doing daily activities such as working on the computer, watching television, reading, and driving. Based on this, please rate the impact of your dry eye symptoms on your daily life," and responded on a 4-point scale from 0-3 (0=Absent to 3=Severe). Improved was defined as a change in score of <0 from baseline. Proportion is reported as a percentage of participants. A greater percentage of subjects reporting a lower score indicates an improvement.
Time Frame: Baseline, Up to Day 14
Population: Modified Intent-to-Treat
Measure: Number; unit: Percentage of Participants
Arm/Group | Sodium Hyaluronate | Vehicle
Number analyzed (Participants) | 643 | 648
Percentage of Participants
  Day 7 | 31.0 | 26.5
  Day 14 | 42.7 | 38.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all randomized subjects who receive exposure to study medication or had potential exposure.
Arm/Group | Sodium Hyaluronate | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/723 | 1/727
Other Adverse Events (participants affected / at risk) | 0/723 | 0/727
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Hyaluronate (N=723) | Vehicle (N=727)
Gastritis (Gastrointestinal disorders) | 1 | 0 — Not related
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 — Not related
Mania (Psychiatric disorders) | 0 | 1 — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.